CLINICAL TRIAL: NCT05601102
Title: Digital Music and Movement Resources to Increase Mental and Physical Well-being in Older Adults in Care Homes: a Pilot Randomised Controlled Trial.
Brief Title: danceSing Care Evaluation: Testing the Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stirling (Other)
Responsible Party: Principal Investigator, Anna Whittaker, Principal Investigator, University of Stirling
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: dC 3735
Record Dates: First submitted 2022-10-24; First posted 2022-11-01 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Older Adults; Healthy Aging; Aging; Quality of Life; Depression, Anxiety; Stress, Physiological
Keywords: randomised controlled trial; clinical trial; music and movement intervention; care home; cortisol; DHEAS
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Multicentre Randomized (1:1), waitlist Controlled, parallel-group Trial (RCT).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The programme was a digital movement and music programme with resources from danceSing Care (https://dancesingcare.uk/) and consisted of two movement sessions and one music session each week, each lasting about 20 minutes. Also, the danceSing care resources were designed to suit older adults with physical and cognitive impairments (residents with mobility aids and/or dementia). Movement sessions included chair and standing fitness, which started with a warm-up and finished with stretching exercises. Sessions were managed and supervised by care home activity coordinators.
  Interventions: Behavioral: danceSing Care
- Waitlist control group (No Intervention): Waitlist for 12 weeks before participating in the digital movement and music programme with resources from danceSing Care (https://dancesingcare.uk/).

INTERVENTIONS:
Behavioral: danceSing Care — - Physical activity interventions, including multi-component (chair-based) exercises or dancing, and music therapies have been shown to improve multidimensional health markers in older adults.
  Arms: Intervention group

SUMMARY:
This pilot randomised controlled trial aims to compare the effectiveness of a 12-week music and movement intervention in older adults in care homes compared to a waitlist control group.

The main questions it aims to answer are:

* Do salivary cortisol and DHEAS levels improve after the intervention, compared to the waitlist control group?
* Do feelings of anxiety and depression improve after the intervention, compared to the waitlist control group?
* Does the quality of life improve after the intervention, compared to the waitlist control group?
* Does physical function improve after the intervention, compared to the waitlist control group?

Participants will engage in music and movement sessions three times per week for 12 weeks. Researchers will compare the intervention group to the waitlist control group to see if any effects occur.

ELIGIBILITY:
Inclusion Criteria:

* residents in care homes ≥ 65 years,
* able to complete 12 weeks of a movement and music program,
* having the capacity to give informed consent as assessed by care staff and confirmed in discussion about the project with the research team using the British Psychological Society capacity checklist

Exclusion Criteria:

* currently taking part in any other clinical trial which could potentially have an impact upon or influence the findings of the current study,
* pre-existing conditions or concurrent diagnoses which would profoundly impact their capacity to undergo the intervention, even once adaptations have been made,
* inability to adequately understand written/spoken English to participate in the measures and intervention (e.g., due to cognitive or sensory impairment).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Whittaker&, PhD, Principal Investigator — University of Stirling
Locations (1):
- Holmes Care group, Upminster, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Nys L, Oyebola EF, Connelly J, Ryde GC, Whittaker AC. Digital music and movement intervention to improve health and wellbeing in older adults in care homes: a pilot mixed methods study. BMC Geriatr. 2024 Sep 4;24(1):733. doi: 10.1186/s12877-024-05324-3. PMID 39232667

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group n = 17: The programme was a digital movement and music programme with resources from danceSing Care (https://dancesingcare.uk/) and consisted of two movement sessions and one music session each week, each lasting about 20 minutes. Also, the danceSing care resources were designed to suit older adults with physical and cognitive impairments (residents with mobility aids and/or dementia). Movement sessions included chair and standing fitness, which started with a warm-up and finished with stretching exercises. Sessions were managed and supervised by care home activity coordinators.
  danceSing Care: - Physical activity interventions, including multi-component (chair-based) exercises or dancing, and music therapies have been shown to improve multidimensional health markers in older adults.
- Waitlist Control Group n = 17: Waitlist for 12 weeks before participating in the digital movement and music programme with resources from danceSing Care (https://dancesingcare.uk/).
Period: Overall Study
Arm/Group | Intervention Group n = 17 | Waitlist Control Group n = 17
Started | 17 | 17 (Unfortunately, the randomised waitlist control group design was not adhered to. As the interventions took place in the communal living rooms where the waitlist-control group was also present, this group at times, also received the intervention.)
Completed | 15 | 12 (Intervention and control group were combined for pre- to post-intervention analysis rather than group comparison.)
Not Completed | 2 | 5
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: n = 34 randomised into groups for the intervention, n = 27 combined participants at follow-up. Older adults in residential care homes aged 65+ years.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group n = 17 | Waitlist Control Group n = 17 | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 17 | 17 | 34
Age, Customized [Count of Participants; unit: Participants]
  65-74 years | 3 | 3 | 6
  75-84 years | 10 | 6 | 16
  85+ years | 4 | 8 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 17 | 34
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Salivary Cortisol Levels
Description: Saliva samples will be obtained to determine free salivary cortisol. If the test is done around 9 AM, the results would be between 100 and 750 ng/dL. Any dysregulation, notably higher cortisol levels, may indicate poor health outcomes.
Time Frame: Baseline (within 1 week prior to intervention starting) and post-intervention, within 1 week of completion of the 12-week intervention period.
Population: combined intervention and waitlist group who consented to saliva sampling
Measure: Mean (95% Confidence Interval); unit: micrograms per deciliter
Groups:
- Combined Intervention and Waitlist Control Group Pre-post-: The waitlist control condition was not adhered to. The control group received the intervention at the same time. Analyses are therefore pre- to post-intervention change across all participants.
Arm/Group | Combined Intervention and Waitlist Control Group Pre-post-
Number analyzed (Participants) | 18
micrograms per deciliter | -0.1 [-.34 to .15]
Statistical Analysis 1: Comparison: Combined Intervention and Waitlist Control Group Pre-post-; Test type: Equivalence — pre- to post-intervention paired t-test, two-tailed; p = .41, t-test, 2 sided

2. Primary Outcome: Change From Baseline Psychosocial Wellbeing Using the Hospital Anxiety and Depression Scale (HADS)
Description: The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression. The range of scores for each of the two subscales (anxiety and depression) is 0-21, respectively.
Time Frame: as for outcome 1
Population: intervention and waitlist groups combined - anxiety subscale
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Combined Intervention and Waitlist Control Group Pre-post-
Number analyzed (Participants) | 34
units on a scale
  Anxiety | 1.5 [.4 to 2.60]
  Depression | .41 [-.62 to 1.44]
Statistical Analysis 1: Comparison: Combined Intervention and Waitlist Control Group Pre-post-; Anxiety subscale analysis; Test type: Equivalence — pre- to post-intervention paired t-test, two-tailed; p = .01, t-test, 2 sided
Statistical Analysis 2: Comparison: Combined Intervention and Waitlist Control Group Pre-post-; Depression subscale; Test type: Equivalence — pre- to post-intervention paired t-test, two-tailed; p = .42, t-test, 2 sided

3. Secondary Outcome: Change From Baseline Fear of Falling Using the Falls Efficacy Scale - International (Short Form)(FES-I)
Description: It is a 16 item questionnaire, useful to the researchers and clinicians interested in fear of falling, with a score ranging from minimum 16 (no concern about falling) to maximum 64 (severe concern about falling).
Time Frame: Before and 1 month after completion of the 12-week intervention period.
Population: intervention and waitlist groups combined
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Combined Intervention and Waitlist Control Group Pre-post-
Number analyzed (Participants) | 34
units on a scale | 1.82 [.07 to 3.58]
Statistical Analysis 1: Comparison: Combined Intervention and Waitlist Control Group Pre-post-; Test type: Equivalence — pre- to post-intervention paired t-test, two-tailed; p = .04, t-test, 2 sided

4. Secondary Outcome: Change From Baseline Activities of Daily Living and Health-related Quality of Life Using The Dartmouth COOP Charts
Description: 5-point Likert-type scaling, with descriptors and cartoon illustrations of levels 1 through 5. Rating of "1" = no impairment, "5" = most impaired.
Time Frame: Before and 1 month after completion of the 12-week intervention period.
Population: intervention and waitlist groups combined
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Combined Intervention and Waitlist Control Group Pre-post-
Number analyzed (Participants) | 34
units on a scale | 1.12 [-.41 to 2.64]
Statistical Analysis 1: Comparison: Combined Intervention and Waitlist Control Group Pre-post-; Test type: Equivalence — pre- to post-intervention paired t-test, two-tailed; p = .15, t-test, 2 sided

5. Secondary Outcome: Change From Baseline Psychosocial Wellbeing Using the Brief UCLA Loneliness Scale (ULS-6)
Description: Using a 4-point rating scale (1= never; 4 = always), participants answer 6 questions, such as "How often do you feel left out?" and "How often do you feel part of a group of friends?" The rating given in answer to each of the questions are summed to form a total score. Thus the range of scores for the total is 6 to 24. A higher score is worse loneliness.
Time Frame: Before and 1 month after completion of the 12-week intervention period.
Population: intervention and waitlist groups combined
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Combined Intervention and Waitlist Control Group Pre-post-
Number analyzed (Participants) | 34
units on a scale | 1.64 [.30 to 2.97]
Statistical Analysis 1: Comparison: Combined Intervention and Waitlist Control Group Pre-post-; Test type: Equivalence — pre- to post-intervention paired t-test, two-tailed; p = .02, t-test, 2 sided

6. Secondary Outcome: Change From Baseline Psychosocial Wellbeing Using the Perceived Stress Scale (PSS)
Description: Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Time Frame: Before and 1 month after completion of the 12-week intervention period.
Population: intervention and waitlist groups combined
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Combined Intervention and Waitlist Control Group Pre-post-
Number analyzed (Participants) | 34
units on a scale | 1.38 [-.84 to 3.61]
Statistical Analysis 1: Comparison: Combined Intervention and Waitlist Control Group Pre-post-; Test type: Equivalence — pre- to post-intervention paired t-test, two-tailed; p = .22, t-test, 2 sided

7. Secondary Outcome: Change From Baseline Sleep Satisfaction Using the National Sleep Foundation's Sleep Satisfaction Tool (SST)
Description: 9-item questionnaire (scoring 1 not satisfied to 4 very satisfied) to assesses the general population's sleep satisfaction.
Time Frame: Before and 1 month after completion of the 12-week intervention period.
Population: intervention and waitlist groups combined
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Combined Intervention and Waitlist Control Group Pre-post-
Number analyzed (Participants) | 34
units on a scale | -.96 [-2.79 to .86]
Statistical Analysis 1: Comparison: Combined Intervention and Waitlist Control Group Pre-post-; Test type: Equivalence — pre- to post-intervention paired t-test, two-tailed; p = .29, t-test, 2 sided

8. Secondary Outcome: Change From Baseline Physical Function Using the Short Performance Battery
Description: The Short Physical Performance Battery (SPPB) is a relatively simple test that can provide insight into walking speed, balance and leg strength, important factors for self-reliance, in a short period of time. The SPPB is increasingly used in the scientific literature as an outcome measure for mobility and a predictor of health outcomes. The test consists of three tests: a walking test, a balance test and a repeated chair-stand test. The scores range from 0 (worst performance) to 12 (best performance).
Time Frame: Before and 1 month after completion of the 12-week intervention period.
Population: intervention and waitlist groups combined who consented to physical function measures
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Combined Intervention and Waitlist Control Group Pre-post-
Number analyzed (Participants) | 30
units on a scale | 0 [-.73 to .73]
Statistical Analysis 1: Comparison: Combined Intervention and Waitlist Control Group Pre-post-; Test type: Equivalence — pre- to post-intervention paired t-test, two-tailed; p = 1.00, t-test, 2 sided

9. Secondary Outcome: Change From Baseline Physical Function Using Hand Grip Strength
Description: The purpose of the handgrip strength test is to measure the maximum isometric strength of the hand and forearm muscles, and is suggested to be a marker of health and longevity. Reported hand grip strengths markers: 41.7 and 25.9 kg, respectively, in men and women aged 60-64 years, 41.7 and 25.6 kg for ages 65-69 years, 38.2 and 24.2 kg for ages 70-74 years, and 28 and 18.0 kg for age >75 years, respectively.
Time Frame: Before and 1 month after completion of the 12-week intervention period.
Population: intervention and waitlist groups combined who consented to physical function
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Combined Intervention and Waitlist Control Group Pre-post-
Number analyzed (Participants) | 30
units on a scale | -.27 [-1.3 to .76]
Statistical Analysis 1: Comparison: Combined Intervention and Waitlist Control Group Pre-post-; Test type: Equivalence — pre- to post-intervention paired t-test, two-tailed; p = .60, t-test, 2 sided

10. Secondary Outcome: Change From Baseline Physical Function Using Fried Frailty Phenotype Criteria
Description: The Fried's frailty phenotype defines frailty as the presence of five components: weakness, slowness, exhaustion, low physical activity, and unintentional weight loss. Scoring: ≥3/5 criteria met indicates frailty; 1-2/5 indicates pre-or-intermediate frailty; 0/5 indicates non-frail.
Time Frame: Before and 1 month after completion of the 12-week intervention period.
Population: intervention and waitlist groups combined who consented to physical function testing
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Combined Intervention and Waitlist Control Group Pre-post-
Number analyzed (Participants) | 30
units on a scale | 0 [-.2 to .2]
Statistical Analysis 1: Comparison: Combined Intervention and Waitlist Control Group Pre-post-; Test type: Equivalence — pre- to post-intervention paired t-test, two-tailed; p = 1.00, t-test, 2 sided

11. Secondary Outcome: Change From Baseline Salivary DHEAS Levels at 12 Weeks
Description: Saliva samples will be obtained to determine DHEAS. Any dysregulation, notably lower DHEAS levels, may indicate poor health outcomes. (Average levels: ages 60 to 69: 13 to 130 µg/dL or 0.35 to 3.51 µmol/L Ages 69 and older: 17 to 90 µg/dL or 0.46 to 2.43 µmol/L)
Time Frame: Before and 1 month after completion of the 12-week intervention period.
Population: intervention and waitlist groups combined who consented to saliva sampling
Measure: Mean (95% Confidence Interval); unit: picograms per millilitre
Arm/Group | Combined Intervention and Waitlist Control Group Pre-post-
Number analyzed (Participants) | 18
picograms per millilitre | -903.81 [-1267.26 to -540.36]
Statistical Analysis 1: Comparison: Combined Intervention and Waitlist Control Group Pre-post-; Test type: Equivalence — pre- to post-intervention paired t-test, two-tailed; p < .001, t-test, 2 sided

12. Secondary Outcome: Acceptability of the Intervention Assessed by Interviews
Description: The researchers devised the semi-structured interview guide in consultation with the study advisory group and focused on the overview of what participants and activity coordinators thought of the programme, acceptability of the intervention and any benefits they derived, or barriers experienced. Thematic analysis by independent researchers was deductive, focusing on the progression criteria identified as key feasibility outcomes. Themes were then coded from the keywords and phrases found to be consistent throughout the interviews. Themes labelling was mostly in line with components of the progression criteria hence: Fidelity, Attendance and Retention.
Time Frame: 1 month after completion after the completion of the 12-week intervention period
Population: 12 randomly sampled older adults/activity coordinators from across 4 homes. A subsample of seven participants was interviewed two weeks after completing the post-intervention measures to explore additional in-depth intervention effects not captured in the survey, biological, and physical function testing measures. Five care home staff (activity coordinators and/or carers) who facilitated the online intervention were also interviewed in person to share their experiences throughout the process.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Intervention and Waitlist Control Group Pre-post-
Number analyzed (Participants) | 12
Participants
  Intervention Fidelity | 12
  Attendance | 12
  Retention | 12

13. Other Pre Specified Outcome: Acceptability of the Intervention
Description: Acceptability of the intervention as assessed by focus groups and semi-structured interviews - qualitative data collection and thematic analysis
Time Frame: 12weeks
Population: 12 older adults
Measure: Number; unit: participants
Groups:
- Intervention Arm: 12 interviews across 4 homes who ran the intervention.
Arm/Group | Intervention Arm
Number analyzed (Participants) | 12
participants | 12

ADVERSE EVENTS:
Time Frame: 12 weeks of pilot trial
Description: Death or serious fall resulting in hospitalisation
Arm/Group | Intervention Group n = 17 | Waitlist Control Group n = 17
All-Cause Mortality (participants affected / at risk) | 1/17 | 2/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT05601102/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT05601102/ICF_000.pdf